CLINICAL TRIAL: NCT02024841
Title: Feasibility Study of Intraperitoneal Docetaxel Combined With Intravenous Cisplatin and Oral TS-ONE for Gastric Cancer Patients With Peritoneal Carcinomatosis
Brief Title: Intraperitoneal Docetaxel With Cisplatin and TS-ONE for Gastric Cancer With Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Lam Ka On, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKUGCDTC01
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
Keywords: Gastric cancer; Peritoneal carcinomatosis; Intraperitoneal docetaxel; Cisplatin; TS-ONE
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraperitoneal docetaxel (Experimental): Intraperitoneal docetaxel in 1litre normal saline infused over 1 hour on day 1 every 3 weeks:
  - Level I: 40mg/m2; Level II: 50mg/m2; Level III: 60mg/m2
  Intravenous cisplatin: 60mg/m2 on day 1 every 3 weeks
  Oral TS-ONE: 40-60mg twice daily on day 1 -14 every 3 weeks
  Interventions: Drug: Intraperitoneal docetaxel

INTERVENTIONS:
Drug: Intraperitoneal docetaxel — Intraperitoneal docetaxel, intravenous cisplatin and oral TS-ONE every 3 weeks for 3 cycles then stop
  Other Names: Intraperitoneal taxotere

SUMMARY:
Phase I study on the maximum tolerated dose (MTD) and the recommended dose (RD) of intraperitoneal docetaxel combined with intravenous cisplatin and oral TS-ONE in gastric cancer patients with peritoneal carcinomatosis

DETAILED DESCRIPTION:
Peritoneal carcinomatosis (PC) is common in advanced gastric cancer, and it carries a poor prognosis; the median survival time is 3 to 6 months. Gastric cancer with PC is considered incurable and patients are subjected to non-surgical treatment, mainly chemotherapy. Currently, there is no established standard treatment for these patients.

Multidisciplinary approach to the treatment of gastric cancer including chemotherapy, radiotherapy and surgery has been developed and survival benefit has been demonstrated in the adjuvant setting. Novel chemotherapeutic agents: taxanes (paclitaxel and docetaxel), irinotecan, oxaliplatin, fluoropyrimidine (TS-ONE and capecitabine) have shown activity in gastric cancer. Various combination chemotherapy regimens for unresectable and metastatic gastric cancer are practised in different parts of the world. Epirubicin, cisplatin and 5-fluorouracil (ECF) are used in Europe, while TS-ONE and cisplatin are commonly used in Asian countries such as Japan and Korea. The median survival time (MST) with these regimens was 8.9 and 13 months, respectively. Use of docetaxel, cisplatin and 5-fluorouracil (DCF) was proposed in the V325 study, MST was 9.2 months but the toxicity (grade 3-4 neutropenia) was reported to be significantly higher in DCF group when compared with CF group. However, there are few trials to study the specific efficacy of these regimens on PC.

Systemic chemotherapy is considered to be less effective against PC due to the existence of the blood-peritoneal barrier (BPB). The barrier inhibits the movement of drugs from systemic circulation to the peritoneal cavity. Intraperitoneal (IP) chemotherapy has the advantage of maintaining a high drug concentration in the peritoneal cavity, and reduces the systemic toxicity. Paclitaxel and docetaxel have been shown to have high peritoneal concentration in animal studies and are considered ideal drugs for IP administration.

Neoadjuvant intraperitoneal/systemic chemotherapy (NIPS) is a new bidirectional induction chemotherapy for treatment of PC from gastric cancer. The aim of NIPS is to induce a reduction of PC volume. Bidirectional means that NIPS could attack PC from both the peritoneal cavity and the subperitoneal blood vessels. Patients with good response to NIPS may undergo subsequent gastrectomy. The use of TS-ONE and IP taxane (paclitaxel/docetaxel) had been studied in phase I and II trials. Ischigami et al. reported 1-year survival rate of 78% and overall response rate of 56% using weekly intravenous and IP paclitaxel combined with TS-ONE. Fujiwara et al. reported 78% patients had negative peritoneal cytology after NIPS and 16 out of 18 patients (88.9%) underwent subsequent gastrectomy, with a MST of 24.6 months. No treatment-related mortality has been reported.

Systemic DCF is associated with significant toxicity, yet it is superior to CF alone in terms of survival (9.2 months vs. 8.6 months, p<0.02). Grade III/IV neutropenia was reported to be 82%. It is postulated that switching from intravenous docetaxel to IP docetaxel may improve its efficacy against PC and reduce the systemic toxicity. TS-ONE contains tegafur, 5-chloro-2,4-dihydroxypyridine (CDHP) and potassium oxonate (Oxo). Dihydropyrimidine dehydrogenase (DPD), which is found in liver, rapidly degrades 5-FU. The presence of CDHP, a specific inhibitor of DPD, allows a high intraperitoneal drug concentration after oral administration of TS-ONE that has been demonstrated in an experimental model.

Therefore we propose a modification of the DCF regimen using IP docetaxel, intravenous cisplatin and oral TS-ONE in the treatment of gastric cancer patients with PC. We aim to study the maximum tolerated dose (MTD) and the recommended dose (RD) of IP docetaxel while using fixed doses of cisplatin and TS-ONE. Data on treatment efficacy will also be recorded. By far there is no study on IP chemotherapy in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Histologic confirmation of gastric adenocarcinoma
* Positive peritoneal cytology or histological proven PC
* Absence of other distant metastases except peritoneum and lymph node(s)
* Adequate bone marrow and organ functions as defined below:
* Leucocyte ≥3.00 x 109/L
* Absolute neutrophil counts ≥ 1.50 x 109/L
* Platelet ≥ 100 x 109/L
* Total bilirubin ≤2 x ULN
* AST/ALT ≤2.5 x ULN
* Creatinine clearance ≥60ml/min
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subjects of child-bearing potential must agree to contraception from screening to 6 months after completion of treatment
* Provision of written informed consent

Exclusion Criteria:

* Any prior anti-cancer therapy for gastric cancer
* Previous exposure to taxane, fluoropyrimidine or platinum chemotherapy
* Previous radiotherapy to abdomen or pelvic region
* Known hypersensitivity to study medication
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Any prior or synchronous malignancy, except,
* Malignancy treated with curative intent and with no evidence of disease for ≥5 years prior to enrollment and considered to be at low risk for recurrence by the treating physician
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Subject is pregnant or breast feeding
* Any serious concomitant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended dose | 2 years

SECONDARY OUTCOMES:
Clinical response rate | 12 weeks
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ka-On Lam, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No